CLINICAL TRIAL: NCT01139398
Title: Effect of Dietary Supplement Limicol on LDL-cholesterol Levels in Moderate Hypercholesterolaemia
Brief Title: Effect of Limicol on (LDL)-Cholesterol Levels in Moderate Hypercholesterolaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L2009-06
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Delivery of Health Care
Keywords: Cholesterol; LDL-cholesterol; Coronary artery disease; Red yeast rice; Plants extract; Cholesterol excess.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Limicol (plant extract) — Artichoke extract, anti-caking agents: dicalcium phosphate, calcium citrate, vegetable magnesium stearate, red yeast rice, microcrystalline cellulose, natural vitamin E, garlic extract, sugar cane policosanols, inositol hexanicotinate, vitamin B3, vitamin B2.
  Other Names: Limicol

SUMMARY:
The purpose of this study is to validate the effectiveness of food supplement Limicol on reducing LDL-cholesterol in moderate hypercholesterolemic volunteers.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), foremost among which ischemic heart disease and stroke, are the leading cause of mortality and morbidity in France. These diseases are multifactorial origin and even if it is not possible to act on risk markers such as age, sex, or heredity, risk factors like high cholesterol, smoking , hypertension, obesity, diabetes and physical inactivity, are the main target of prevention strategies.The dydlipidémies have a role in the formation of CVD in participating in the genesis of atherosclerosis. The cholesterol and LDL-cholesterol in particular is subject to oxidation process in plasma. The molecules of oxidized LDL-cholesterol, small and dense, easily penetrate the arterial endothelial wall and are greeted by macrophages. Following a succession of different processes including inflammation, atherosclerotic plaque is formed. The result is either an arteriopathy when the arterial lumen narrowing, or atherothrombosis in the event of plaque rupture. Given this pathophysiology, reduce blood lipids, including LDL-cholesterol and reducing oxidation and inflammation are interesting strategies in the context of cardiovascular prevention. Several scientific study showed that nutritional supplementation with some plant extracts such as artichokes, garlic, red yeast rice, or the sugar cane policosanol helps to reduce several cardiovascular risk factors including regulate concentrations of circulating lipids.

The objective of this study is to validate the effectiveness of Limicol, formulated with proven scientific data on the reduction of LDL-cholesterol in volunteers with moderate hypercholesterolaemia (LDL-cholesterol).

ELIGIBILITY:
Inclusion Criteria:

* About 18 to 65 years (inclusive).
* Subject has a stable weight for at least three months before the start of the study.
* Subject able and willing to comply with the protocol and agreeing to give their consent in writing.
* Subject affiliated with a social security scheme.
* Subject willing to be included in the national register of volunteers who lend themselves to biomedical research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol levels | 4 months

SECONDARY OUTCOMES:
Total cholesterol, HDL-cholesterol, triglycerides levels | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Nantes, France